CLINICAL TRIAL: NCT03484208
Title: Evaluation of a Fracture Liaison Service in the Osteoporosis Care
Status: Terminated | Type: Observational
Why Stopped: PI's choice
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: FILIERE FRACTURE
Record Dates: First submitted 2018-03-25; First posted 2018-03-30 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Osteoporotic Fractures
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: osteoporotic fracture liaison service — a specific nurse calls patient and propose them to follow the osteoporotic fracture liaison service

SUMMARY:
The St JOSEPH'S HOSPITAL set up a fracture liaison service for osteopotic fracture. A specific nurse screens eligible patient admitted in emergency yard and call them to propose a bone densitometry and a medical coverage..

The aim of the study is to evaluate this new organisation

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 95 years old.
* Admitted in emergency yard for law energy trauma

Exclusion Criteria:

* feet fracture
* fracture on prothesis
* patient transferred elsewhere
* homeless people
* patient with lot of comorbidities

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in emergency yard for low energy fracture
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
valuable osteoporosis care | Month 1
  valuable osteoporosis care means a bone densitometry for minor fracture and a medical treatment for major fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France